CLINICAL TRIAL: NCT00682487
Title: Hair Cortisol and the Risk of Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Dr David Pereg, Department of Internal Medicine A and Cardiology devision, Meir Medical Center
Other Study IDs: 0246-07-MMC
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2009-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Myocardial infarction; Stress; Hair Cortisol
MeSH Terms: conditions — Myocardial Infarction | interventions — Hydrocortisone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: patients admitted to the cardiology department with acute Myocardial infarction.
  Interventions: Other: Hair sampling for cortisol
- 2: patients admitted to an internal medicine department due to reasons other than an acute thrombotic event
  Interventions: Other: Hair sampling for cortisol

INTERVENTIONS:
Other: Hair sampling for cortisol — Hair sampling for cortisol
  Groups: 1
Other: Hair sampling for cortisol — Hair sampling for cortisol
  Groups: 2

SUMMARY:
Aim of the study:

To evaluate whether hair cortisol levels are elevated in patients admitted with acute MI compared to controls.

Study steps:

1. Introduction of the study to the participants and inform consent signing
2. Collection of clinical and demographic data
3. Scalp hair sampling- samples will be sent for laboratory analysis
4. Analysis of the results

DETAILED DESCRIPTION:
Acute physical stressors such as surgery, trauma and intense physical exertion are well-known triggers of cardiovascular events. The connection between acute emotional stress and the heart has been controversial for many years. However, emotional stressors are now increasingly recognized as precipitants of cardiovascular events including myocardial infarction (MI). For example, on the day of the Los Angeles earthquake in 1994 the number of cardiac deaths and hospital admissions for acute myocardial infarction was 2-5 times higher than the usual rate. Furthermore, the risk of myocardial infarction in the short period following an acute emotional stress such as anger outburst, seems to be twice that of other periods and may be a more common precipitant than physical exertion1. While the association between acute stress and cardiovascular mortality and morbidity is well established, controversy still exists whether there is the same association with chronic stress, both physical and emotional. Data regarding this question are extremely limited since there has been no objective and reliable mode for the assessment of physical stress and for the quantification of overall chronic stress. Furthermore, the fact that all the information regarding the association between chronic stress and acute MI derives from retrospective studies further complicates this issue.

Both physical and emotional stress activate several neuroendocrine systems, the most important being the hypothalamic-pituitary-adrenal axis that stimulates the production and secretion of glucocorticoids (especially cortisol) from the adrenal cortex. Therefore, cortisol is considered to be a "stress hormone" and higher levels of serum cortisol have been observed in patients with acute stress such as those presented with acute MI, compared to healthy controls.

Currently, there are several modalities for measuring cortisol levels including serum, urinary and salivary techniques. However, all these methods represent indicators of acute stress and do not reflect accumulation of stress over time.

Recently there has been a growing interest in measuring hair cortisol level. Hair grows approximately 1 centimeter per month, and hair analysis accurately reflects long-term endogenous production of cortisol. This provides for the first time a reliable mode for the measurement of the accumulation of cortisol over time and a potential biomarker of chronic stress. Indeed, several reports have demonstrated an association between high hair cortisol levels and chronic stress in both animal models and in humans. Nevertheless, the possible association between hair cortisol and the risk of acute MI has not been studied yet.

Aim of the study:

To evaluate whether hair cortisol levels are elevated in patients admitted with acute MI compared to controls.

ELIGIBILITY:
Inclusion Criteria:

1. Cases- patients with acute MI ( elevated cardiac enzymes + chest pain or typical ECG changes)
2. Controls- patients admitted to an internal medicine department due to reasons other than acute MI or stroke.

Exclusion Criteria:

1. Corticosteroid treatment in the last 12 months
2. Diagnosis or Cushing's or Addison's disease
3. Treatment with hormone replacement therapy
4. Treatment with oral contraceptives
5. Colored heir
6. Inability to sign inform consent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases: Patients admitted to the cardiology department due to acute myocardial infarction Controls: Patiens admitted ro an Internal Medicine department due to non-thrombotic disease.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
hair cortisol levels in patients admitted with acute MI compared to controls | at enrollment

SECONDARY OUTCOMES:
the association between hair cortisol levels and the prognosis of patients with acute MI. | at enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Brotman DJ, Golden SH, Wittstein IS. The cardiovascular toll of stress. Lancet. 2007 Sep 22;370(9592):1089-100. doi: 10.1016/S0140-6736(07)61305-1. PMID 17822755
- [Background] Yamada J, Stevens B, de Silva N, Gibbins S, Beyene J, Taddio A, Newman C, Koren G. Hair cortisol as a potential biologic marker of chronic stress in hospitalized neonates. Neonatology. 2007;92(1):42-9. doi: 10.1159/000100085. Epub 2007 Mar 14. PMID 17356304
- [Background] Sauve B, Koren G, Walsh G, Tokmakejian S, Van Uum SH. Measurement of cortisol in human hair as a biomarker of systemic exposure. Clin Invest Med. 2007;30(5):E183-91. doi: 10.25011/cim.v30i5.2894. PMID 17892760
- [Background] Kalra S, Einarson A, Karaskov T, Van Uum S, Koren G. The relationship between stress and hair cortisol in healthy pregnant women. Clin Invest Med. 2007;30(2):E103-7. doi: 10.25011/cim.v30i2.986. PMID 17716540
- [Background] Davenport MD, Tiefenbacher S, Lutz CK, Novak MA, Meyer JS. Analysis of endogenous cortisol concentrations in the hair of rhesus macaques. Gen Comp Endocrinol. 2006 Jul;147(3):255-61. doi: 10.1016/j.ygcen.2006.01.005. Epub 2006 Feb 17. PMID 16483573